CLINICAL TRIAL: NCT06700473
Title: Effects of Reiki Intervention During Labor on Pain, Fear, and Birth Experience in Primiparous Women: A Randomized Controlled Trial
Brief Title: Effects of Reiki Intervention During Labor on Pain, Fear, and Birth Experience
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Ozlem TAS, PhD Candidate, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024/303
Record Dates: First submitted 2024-11-20; First posted 2024-11-22 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Labour
Keywords: Reiki, Labour Pain, Delivery, Birth Experience, Fear
MeSH Terms: conditions — Labor Pain | interventions — Therapeutic Touch

STUDY DESIGN:
Intervention Model Description: Single-Blind Randomized Controlled Trial
Who Masked: Participant
Masking Description: After being randomized as experimental and control groups, primiparous pregnant women will be prevented from interacting with each other in order not to be affected by the interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reiki (Experimental): Before the intervention, when their cervical dilatation is 4-5 cm, EC-1, EC-2 and EC-3 will be applied to pregnant women in all groups. After the initial data collection, the researcher TC will apply reiki for approximately 15-20 minutes to pregnant women in the reiki group with cervical dilatation of 4-5 cm. Immediately after the first intervention, the second EC-2 and EC-3 measurements will be performed. The third EC-2 and EC-3 measurements will be performed when the cervical dilatation is 6-7 cm and then the fourth EC-2 and EC-3 measurements will be performed after 15 minutes of reiki application. The fifth EC-2 and EC-3 measurements will be performed when the cervical dilatation is 8-9 cm, followed by 15 minutes of reiki and the sixth EC-2 and EC-3 measurements. The final data will be collected one hour after delivery of the placenta with the seventh VAS measurement and EK-4. The EC-4 will also be re-evaluated by the researchers online at the sixth postpartum week.
  Interventions: Other: reiki
- Control (No Intervention): Pregnant women in the control group will receive routine midwifery care during labor. Both groups will not receive any non-pharmacologic intervention for pain management. All women will receive one-to-one support from midwives during labor.

INTERVENTIONS:
Other: reiki — Before the intervention, when their cervical dilatation is 4-5 cm, EC-1, EC-2 and EC-3 will be applied to pregnant women in all groups. After the initial data collection, the researcher TC will apply reiki for approximately 15-20 minutes to pregnant women in the reiki group with cervical dilatation of 4-5 cm. Immediately after the first intervention, the second EC-2 and EC-3 measurements will be performed. The third EC-2 and EC-3 measurements will be performed when the cervical dilatation is 6-7 cm and then the fourth EC-2 and EC-3 measurements will be performed after 15 minutes of reiki application. The fifth EC-2 and EC-3 measurements will be performed when the cervical dilatation is 8-9 cm, followed by 15 minutes of reiki and the sixth EC-2 and EC-3 measurements. The final data will be collected one hour after delivery of the placenta with a seventh VAS measurement and administration of the EC-4. The EC-4 will also be reassessed by the researchers online at six weeks postpartum
  Arms: Reiki

SUMMARY:
Childbirth is an important and often stressful experience for many women, and labor pain is common among women. While labor pain is a natural part of the birth process, its severity and management can have a significant impact on an expectant mother's overall health and birth experience. Studies examining the effects of Reiki on alleviating the pain and fear experienced by pregnant women during labor are limited. In this context, understanding the effects of Reiki practices in the birth process may be important for both clinical practice and future research.

DETAILED DESCRIPTION:
Failure to control pain can cause the mother to experience fear and stress, which can increase the risk of complications during labor and indirectly have negative effects on the newborn. There is a strong association between labor pain and fear. Fear can increase the perception and intensity of pain, making the labor process more challenging and difficult to manage. This can negatively affect the mother's overall birth experience and complicate both the physical and emotional aspects of the birth process. A woman's birth experience also has an impact on her birth memory. A positive birth experience can cause a woman to evaluate the birth process as peaceful and satisfying, which positively shapes birth memory. The use of complementary and alternative therapies is increasing every year. Although Reiki has found application in various fields, there is no information in the available literature on its use in the management of labor pain. Reiki is a complementary treatment method based on the "energy approach" and is generally recognized as safe and without side effects.

ELIGIBILITY:
Inclusion Criteria:

Between the ages of 18 and 35, primiparous, singular primarily experiencing pregnancy, without risky pregnancy status (GDM, HT, etc.), during the birth week, literate Speaks and understands Turkish, 4 cm cervical dilatation

-

Exclusion Criteria:

To have attended a childbirth preparation course, Knowledge of coping with labor pain and fear of childbirth during pregnancy, Presence of chronic disease in the mother, Previous uterine surgery, Having become pregnant through assisted reproductive technologies, Hearing problems Being diagnosed with a known serious psychiatric illness.

-

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — women as labor will take place
Enrollment: 54 (Estimated)
Dates: Start 2024-11-02 (Actual); Primary Completion 2025-04-02 (Estimated); Study Completion 2025-05-02 (Estimated)

PRIMARY OUTCOMES:
labour pain | 5 hours
  reduction of labor pain Visual Analog Scale (VAS) (Annex-2): Visual Analog Scale (VAS) is a scale developed by Price et al. in 1983 and used to measure pain intensity and for pain monitoring. The VAS is 10 cm long and the two ends are named differently. On the scale, '0' indicates no pain and '10' indicates the most severe level of pain. VAS is a measurement tool that is frequently and reliably used to assess labor pain (Price et al., 1983; Mutlu & Özkaya, 2021). VAS measurement data will be used to test hypothesis H1. After the primiparous pregnant women included in the study were assigned to the reiki intervention and control groups, the scale will be applied to measure the pretest data when the cervical opening was 4-5 cm before any intervention was applied and to ensure pain equivalence in the groups.

SECONDARY OUTCOMES:
labour fear | 5 hours
  reducing the fear of childbirth Birth Fear Scale (ANNEX-3): The scale was developed by Wijma (2002), and its Turkish validity and reliability was conducted by Serçekuş et al. This scale is designed to assess fear during labor and consists of 10 items. The administration time varies between 30-90 seconds. Participants are asked to give each item a score between 1 (completely disagree) and 10 (completely agree). The minimum score is 10 and the maximum score is 100; a high score indicates a high level of fear. It is very practical to administer. The scale consists of 5 positive (1, 3, 5, 7, 10) and 5 negative (2, 4, 6, 8, 9) items. Positive items are reverse scored. After the primiparous pregnant women included in the study were assigned to the reiki treatment and control groups, EK-2 will be applied during the birth process follow-up. The scale will not be applied in the 1st hour after delivery.
birth memory | 5 hours
  creating positive birth memory Birth memory and recall scale (BMRS) (ANNEX-4): Developed in 2014 by Foley et al. "Birth Memory and Recall Scale," In 2021, it was adapted into Turkish by Topkara and Çağan. The 7-point Likert-type scale consists of 21 items in total and has six different dimensions: "Emotional Memory," 'Ambivalent Emotional Memory,' 'Centrality of Memory,' 'Consistency and Reliving,' 'Sensory Memory' and "Involuntary Recall." The highest score that can be obtained from the scale is 147 and the lowest score is 6. High scores on the Emotional Memory subscale indicate that the mother has more intense negative feelings about the birth experience, while high scores on the Ambivalent Emotional Memory subscale indicate that the mother has more complex and contradictory feelings about the birth experience.

CONTACTS AND LOCATIONS:
Overall Officials: Uncu, Principal Investigator — Istanbul University - Cerrahpasa; Comert, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- İstanbul Eğitim Araştırma Hastanesi, Istanbul, Zeytinburnu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Isbir GG, Sercekus P. The Effects of Intrapartum Supportive Care on Fear of Delivery and Labor Outcomes: A Single-Blind Randomized Controlled Trial. J Nurs Res. 2017 Apr;25(2):112-119. doi: 10.1097/JNR.0000000000000129. PMID 28277391
- See also: https://pubmed.ncbi.nlm.nih.gov/28277391/ — https://pubmed.ncbi.nlm.nih.gov/28277391/
- Available data/document: Individual Participant Data Set: 10.1097/JNR.0000000000000129. — https://pubmed.ncbi.nlm.nih.gov/28277391/ — https://pubmed.ncbi.nlm.nih.gov/28277391/